CLINICAL TRIAL: NCT04334616
Title: Post Operative Sore Throat: Comparison of Macintosh Laryngoscope Versus Video Laryngoscope in Patients Intubated by Anaesthesia Trainee
Brief Title: POST: Comparison of Macintosh Laryngoscope vs Video Laryngoscope in Patients Intubated by Anaesthesia Trainee
Acronym: POST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Amin Ahmed Kapadia, Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4750-Ane-ERC-17
Record Dates: First submitted 2020-03-28; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Sore Throat
Keywords: Video Laryngoscope; Macintosh Laryngocsope; VDL; Karl Storz Video Laryngoscope; Intubation; Post Operative Sore Throat; Anaesthesia Trainee
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial (Observer Blinded)
Who Masked: Participant, Investigator
Masking Description: After approval from Ethical Review Committee potential patients will be screened in the ward. After eligibility, the consent will be administered by the study investigators. If patient agree to participate and signed the consent, he/she will be enrolled in the study. Selected patients will be randomly allocated by a computer-generated number, either into conventional laryngoscopy (CL) group or video laryngoscopy (VDL) group through sealed envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conventional Laryngocope (Active Comparator): Patients in this arm will be intubated with conventional Macintosh laryngoscope
  Interventions: Device: Macintosh Conventional Laryngocope
- Video Laryngocope (Active Comparator): Patient in this arm will be intubated with Karl Storz Video Laryngoscope
  Interventions: Device: Video Laryngocope

INTERVENTIONS:
Device: Video Laryngocope — VDL used for VDL arm
  Arms: Video Laryngocope
Device: Macintosh Conventional Laryngocope — Used for Conventional laryngocope arm
  Other Names: Conventional Laryngocope
  Arms: Conventional Laryngocope

SUMMARY:
OBJECTIVES The objective of this study is to compare the frequency of POST in patients intubated by trainee anaesthetist using Video LaryngoscopeTM(VDL) versus Conventional Macintosh Laryngoscope (CL) at a tertiary care hospital in Karachi, Pakistan

OPERATIONAL DEFINITIONS

1. Sore Throat: A sore throat is pain, scratchiness or irritation of the throat usually from irritation or inflammation of the throat (pharynx)(11).

   The visual analogue scale (0-10) will be used to evaluate the severity of sore throat
2. Trainee Anesthetist: Anesthesia residents level I and II having experience of more than six months. They will have to achieve the initial competence of doing intubation under direct supervision and need to be familiar with conventional as well as VDL technique.

HYPOTHESIS:

NULL HYPOTHESIS: There is no difference in the frequency of POST in patients intubated by trainee anaesthetists using VDLTM versus conventional Macintosh laryngoscope.

ALTERNATE HYPOTHESIS: There is a difference in the frequency of POST in patients intubated by trainee anaesthetists using VDLTM versus conventional Macintosh laryngoscope.

DETAILED DESCRIPTION:
MATERIAL AND METHODS

SETTING: The study will be conducted at main Operating Room, Department of Anaesthesiology, Aga Khan University Hospital Karachi.

DURATION OF STUDY: This study will be conducted for a period of one year or till the completion of sample size after approval of synopsis by ERC and CPSP.

SAMPLE SIZE:

W.H.O software is used to calculate sample size (See Annexure 1) Frequency of POST in VDL group = 28% (7) Frequency of POST in CL Group =54% (7) Power of the test = 80% Type I error= 5% Sample size in each group =55 (Total sample size 110)

STUDY DESIGN:

Randomized Control Trial (Observer Blinded)

SAMPLING TECHNIQUE:

Non probability consecutive sampling

DATA COLLECTION: After approval from Ethical Review Committee potential patients will be screened in the ward. After eligibility, the consent will be administered by the study investigators. If patient agree to participate and signed the consent, he/she will be enrolled in the study. Selected patients will be randomly allocated by a computer-generated number, either into conventional laryngoscopy (CL) group or video laryngoscopy (VDL) group through sealed envelopes. All patients will be managed with general anaesthesia requiring control mode ventilation and intubation. The direct supervision of consultant anesthetist involved in the study protocol would be there for every case. After instituting routine American society of Anaesthesiologist (ASA) recommended monitoring standards, induction of anaesthesia would be done by the consultant anaesthetistwith Propofol 1.5-2 mg/Kg, Nalbuphine 0.1 milligram per Kg and Atracurium 0.5 mg/Kg. The readiness of intubating conditions will be judged by orbicular oculi response of train of four stimuli. Patient would be considered ready to intubate when there will be no response to the neuromuscular stimuli. The head of the patient will be placed in sniffing position with under head pillow to facilitate the sniffing position.Selection of VDL or ML will be done as per consecutive sampling. Patient in Macintosh laryngoscopy group (MLG) are going to be intubated by trainee anaesthetist as defined by operational definition with laryngoscope size 3 or 4 blade as per the decision. Similarly the patient in (VLG) will be intubated by trainee anaesthetist as defined earlier with laryngoscope size 3 or 4 as per decided plan. Intubation will be done by trainee anaesthetist using appropriate size of endotracheal tube (ETT).The size 7-7.5 mm ID would be used for adult females, while male patients will require size 8-8.5 mm ID of ETT. All ETT tubes will be lubricated with water-based gel (Aplicare Lubricating Jelly) before intubation. Number of attempts of Laryngoscopy will be noted along with the time taken if less than or greater than 30 seconds also if any alteration like bougie was used. The inflation of the cuff would be guided by any obvious leak as measured by the APL bag valve pressure of 20 mm Hg. Later on inflation of cuff pressure would also be confirmed by pressure manometer. The cuff pressure between 20-25 mm Hg is said to be adequate. The intubation time including the number of intubation attempts or any other maneuver used to aid the intubation will be noted down. Orogastric tube lubricated by water based gel (Aplicare Lubricating Jelly) will be passed in all patients. Number of attempt in passing Orogastric Tube or if the aid of Magill forceps used will be noted.All patients would be positioned supine initially and then head up (reverse trandelenberg), as per surgeons preference which is usual for laparoscopic general surgical procedures Anesthesia will be maintained with Isoflurane in mixture of O2/Air. Dual antiemetic prophylaxis that is dexamethasone 0.1 mg/Kg at start and Ondansteron 0.1 mg/Kg at the end would be used for every patient. Endotracheal tube cuff pressurewill be regularly checked at 30 mins interval. Patient will be excluded if the duration of surgery exceeds one hundred and fifty minutes. Patient will be reversed from anaesthesia when fully recovered from paralytic effect of Atracurium. This again will be judge by twitch monitoring. All patients will be extubated as guided by the subjective and objective criteria of extubation. Reversal of neuromuscular paralysis will again be assessed by twitch response to train of four stimuli at orbicularis oculi muscle. Patient would be given reversal once all four twitches would be there. Patient would be observed for postoperative sore throat at 1, 12 and 24 hours post operatively by the primary investigator who is blinded to the group allocation. The visual analogue scale (0-10) will be used to evaluate the severity of sore throat. The definite measurement of POST will be taken at 24 hours.

ADVERSE EVENTS MANAGEMENT In investigators opinion, there would be no adverse event related to the trial protocol. However, if any event either serious or non-serious happened then will be reported to the ERC and other relevant entities are per institutional guidelines.

DATA ANALYSIS: All statistical analysis will be performed using statistical packages for social science version 19 (SPSS Inc., Chicago, IL). Mean and standard deviation will be computed for age, weight, height, BMI. Frequency and percentage will be computed for gender, mallampatti grade, Type of Laryngoscope, Alteration of airway management at intubation, Cormack &Lehane intubation grade, Number of attempts of Laryngoscopy and sore throat (at 1 hr., 12 and 24 hrs.). Both groups will be compared by Chi-square test for frequency of POST between both groups, P value ≤0.05 will be considered significant.

Stratification analysis will be performed to observe effect of confounding variables like age, BMI, gender, mallampatti grade, Type of Laryngoscope, Alteration of airway management at intubation, Cormack & Lehane intubation grade, duration of intubation and number of attempts of Laryngoscopy. After stratification Chi-square test will be applied to compare POST between groups. p≤0.05 will be considered significant

DATA MANAGEMENT AND STORAGE Data will be stored in lock and key and no one will access other than study investigators. Electronic data would be password protected. Data will be stored for 15 years as per GCP and other regulatory guidelines. Data will be frequently monitored by PI for quality checks and queries will be resolved timely basis.

ELIGIBILITY:
Inclusion Criteria:

1. All adult patient of age between 20-60 year
2. American society of Anesthesiologist grade I and II
3. Scheduled for elective laparoscopic cholecystectomy
4. Both male and female genders

Exclusion Criteria:

1. Anticipated difficult airway as assessed by limited mouth opening (< 2 finger breadth), Limited neck extension.
2. Obesity having BMI>30 kg/m2
3. Any anatomical air way abnormality like cancers of oropharngeal cavity, patient who got radiotherapy in head and neck region known to the primary investigator through patients history
4. Patient having history of GERD requiring rapid sequence induction with cricoid pressure
5. Duration of the surgery exceeding two and a half hours (150 minutes)
6. Patient not intubated within three laryngoscopy attempt

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Post Operative Sore Throat | 24 hours
  Patient will be observed for postoperative sore throat post operatively by the primary investigator who is blinded to the group allocation. The visual analogue scale (0-10) will be used to evaluate the severity of sore throat. The definite measurement of POST will be taken at 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided